CLINICAL TRIAL: NCT05914246
Title: VIOLA PMS Clinical Protocol
Brief Title: VIOLA Post Market Surveillance Clinical Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Graft Solutions Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD0314
Record Dates: First submitted 2023-05-28; First posted 2023-06-22 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease
Keywords: CABG; Coronary artery bypass grafting
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CABG surgery with use of VIOLA (Experimental): patients will be treated for routine CABG, using VIOLA for maintaining hemostasis during suturing of multiple aortic anastomoses
  Interventions: Device: VIOLA proximal seal

INTERVENTIONS:
Device: VIOLA proximal seal — VIOLA proximal seal system for maintenance of hemostasis when suturing the aortic anastomoses

SUMMARY:
The goal of this post marketing surveillance clinical trial is to learn about VIOLA as a proximal seal device in patients undergoing coronary artery grafting (CABG) surgery. The main objective is to evaluate the clinical safety and performance of the VIOLA. Participants will be treated with routine CABG with use of VIOLA for maintaining hemostasis when suturing the proximal anastomosis. Patients will be followed for any clinical events at 6 weeks and 9 months post surgery.

DETAILED DESCRIPTION:
The goal of this post marketing surveillance clinical trial is to collect post market data on the safety and performance of VIOLA as a proximal seal device in patients undergoing coronary artery grafting (CABG) surgery. The main objective is to evaluate the clinical safety and performance of the VIOLA. Participants will be treated with routine CABG with use of VIOLA for maintaining hemostasis when suturing the proximal anastomosis. Data will be collected intraoperatively, at discharge, at 6 weeks, and at 9 months post CABG.

ELIGIBILITY:
Inclusion Criteria:

1. Patient scheduled for isolated CABG on clinical grounds
2. One or more bypass grafts originating from the aorta
3. Ability to give their informed written consent
4. Ability and willingness to comply with study follow up requirements
5. Patient is ≥ 18 years of age

Exclusion Criteria:

1. Emergency CABG surgery (cardiogenic shock, inotropic pressure support, IABP)
2. Prior clinical stroke less than one year before surgery
3. Pre-operative neurological deficits
4. Chronic atrial fibrillation
5. Aortic external diameter less than 25 mm measured intraoperatively
6. No proximal aortic anastomosis eligible for VIOLA use, assessed intraoperatively according to surgeon's discretion (E.G inadequate punch size, thin-walled aorta).
7. Symptomatic carotid disease
8. Acute MI within 24 hours of planned surgery
9. EuroScore II ≥ 4
10. Known allergy to nickel
11. Women of child bearing age
12. Participating in any other investigational study for either drug or device which can influence collection of valid data under this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Technical success of the VIOLA device | Acute, intraoperative
  Proportion of proximal anastomoses that were completed without use of an aortic clamp

SECONDARY OUTCOMES:
Sealing quality | Acute, intraoperative
  Sealing quality will be assessed by the surgeon using a 3-point Likert scale. Sealing will be assessed as: 1) Perfect; 2)Acceptable; or 3) Unacceptable
Ease of proximal anastomosis suturing | Acute, intraoperative
  Ease of suturing will be assessed by the surgeon using a 5-point Likert scale where 1=Poor and 5=Excellent

CONTACTS AND LOCATIONS:
Overall Officials: Gil Bolotin, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No